CLINICAL TRIAL: NCT00867802
Title: Mindfulness Intervention For Child Abuse Survivors
Brief Title: Mindfulness Intervention For Child Abuse Survivors (MICAS)
Acronym: MICAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Brian Berman, Director of Research Center for Integrative Medicine, University of Maryland, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00041191
Record Dates: First submitted 2008-12-08; First posted 2009-03-24 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Child Abuse Survivors
Keywords: MICAS; MBSR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness- Based Stress Reduction: Active Comparator (Experimental): Mindfulness-Based Stress Reduction program
  Interventions: Behavioral: Mindfulness-Based Stress Reduction program

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction program — Mindfulness- Based Stress Reduction comprising of 8 classes and a one-day retreat, taught over a period of 6 weeks. Intervention also includes practice at home for 20-30 minutes.

SUMMARY:
The purpose of this study is to assess the effect of meditation training called Mindfulness-Based Stress Reduction on reducing the symptoms of psychological distress among adult survivors of child abuse.

DETAILED DESCRIPTION:
The specific aims of the project are:

1. To determine whether Mindfulness- Based Stress Reduction program is associated with a reduction in symptoms of depression, anxiety, and psychological distress.
2. To assess indications of efficacy, assess feasibility of enrollment and compliance among this patient population
3. Provide pilot data that can be used to apply for larger grants to more fully develop this approach

ELIGIBILITY:
Inclusion Criteria:

* A history of child abuse, as attested by the potential participant
* Currently in therapy with a licensed psychotherapist (psychiatrist, psychologist, social worker).
* Plans to remain in therapy with a licensed psychotherapist (psychiatrist, psychologist, social worker) for the duration of the study.
* Recommendation made by the potential participant's licensed psychotherapist (psychiatrist, psychologist, social worker) the Mindfulness-Based Stress Reduction program would be an appropriate adjunct therapy for his or her client.
* Score of 0.50 or higher on the General Severity Index of the Brief Symptom Inventory, indicating psychological distress above the normal population.
* Aged 21 or above.
* Ability to read and write English.
* Able to attend 10 courses and assessment visits over a 6-week period.
* Willing to practice skills for 20-30 minutes per day 6 days a week, during the course.

Exclusion Criteria:

* Major psychiatric illness (bipolar disorder, schizophrenia, dissociative identity disorder, or others).
* Active alcoholism or drug dependency.
* Any psychological or physical illness the investigator feels would prohibit full participation in the course.
* Currently enrolled in another clinical trial.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To administer the Brief Symptom Inventory (BSI) questionnaire at each visit in order to assess psychological distress. | 6 weeks

SECONDARY OUTCOMES:
Trauma Symptom Inventory to all participants at each visit. Administer the Beck Depression Inventory (BDI) to all participants. Functional Assessment of Chronic Illness Therapy spiritual Well-Being (FACIT-SP) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Pradhan, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Kernan Hospital, Baltimore, Maryland, United States